CLINICAL TRIAL: NCT00102271
Title: Evaluation of the Mechanism of NO Formation and Pharmacokinetics of Systemic Nitrite Infusion
Brief Title: Nitrite Infusion Studies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050088; 05-H-0088
Record Dates: First submitted 2005-01-25; First posted 2005-01-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-12

CONDITIONS: Healthy
Keywords: Sodium Nitrite; Oxypurinol; Ascorbic Acid; Hypoxic Gas; Forearm Blood Flow; Healthy Volunteer; HV
MeSH Terms: interventions — Oxypurinol; Sodium Nitrite

INTERVENTIONS:
Drug: Oxypurinol
Drug: Sodium Nitrite

SUMMARY:
This study will examine 1) how nitrite (a natural blood substance that relaxes blood vessels) increases blood flow and lowers blood pressure, and 2) how to increase the effects of nitrite on blood pressure.

Healthy volunteers between 21 and 40 years of age may be eligible for this study. They must be non-smokers and have no history of high blood pressure, high cholesterol, or diabetes. Candidates are screened with a medical history, physical examination, electrocardiogram, and blood tests. This study is either done in the NIH Clinical Center intensive care unit or on the general clinical ward. Participants are enrolled in Part A of the study. After completion of Part A participants will be enrolled in Part B of the study.

Part A:

Participants lie in a reclining chair during the study. Small catheters (plastic tubes) are inserted into an artery and vein in the forearm. Another tube is placed in the vein of the opposite arm. Blood pressure cuffs are placed around the upper arm and wrist, and a strain gauge (a rubber band-like device) is placed around the forearm. This device helps us to measure blood flow through the arm. When the blood pressure cuffs are inflated, blood flows into the forearm, stretching the strain gauge at a rate proportional to the blood flow. Pressure cuffs and a strain gauge are also placed on the other arm. After 20 minutes, blood pressure and blood flow are measured in both forearms. Then blood is drawn from the tube in the right vein to measure blood counts, proteins, and other chemicals. Participants then are given small doses of either saline, ascorbic acid, or a medicine called oxypurinol, a form of a drug that is often taken to prevent gout. After 30 minutes, sodium nitrite is injected in increasing doses into the artery for 30 minutes. Blood flow is measured and blood is drawn every 5 minutes during the infusion. At the end of the 30 minutes, blood is drawn from the vein every 30 minutes for 3 hours. After 3 hours, sodium nitrite infusions are restarted for 2 hours and blood flow is measured and samples collected every 30 minutes during this period.

Part B: Participants lie in a reclining chair during the study. A small catheter (plastic tube) is placed in the artery of the left forearm to draw blood samples. A larger catheter called a central line is placed in a deeper vein in the neck. Another tube is advanced through the central line into the chambers of the heart, through the heart valve, and into the lung artery to measure pressures in the heart and lungs. Blood is drawn after 30 minutes to obtain baseline measurements. Then saline (sterile salt water) is put into the tube in the lung artery. Blood pressure cuffs are placed around the upper arm and wrist, and a strain gauge (a rubber band-like device) is placed around the forearm, which helps us to measure flow through the arm. When the cuffs are inflated, blood flows into the forearm, stretching the strain gauge at a rate proportional to the blood flow. Pressure cuffs and a strain gauge are also placed on the other arm. After 20 minutes, blood pressure and blood flow are measured in the forearm and blood samples are drawn from the tube in the left artery to measure blood counts, proteins, and other chemicals.

Subjects then breathe a mixture of oxygen and nitrogen through a facemask for 30 minutes, then room air for 30 minutes, and then the oxygen and nitrogen mixture for another 30 minutes. While breathing the mixture the second time, sodium nitrite is injected through the tube in the artery in three increasing doses for 5 minutes each. Every 5 minutes during the infusion blood is drawn from the tubes in the neck. Forearm blood flow is also measured every 5 minutes. After 30 minutes, the subject breathes room air for 3 hours and 15 minutes and then the sodium nitrite is injected again in three increasing doses for 5 minutes each. Every 5 minutes during the infusion blood is taken from the tube in the neck and forearm blood flow is measured

DETAILED DESCRIPTION:
Although regional synthesis of nitric oxide (NO) by the endothelium contributes importantly to local vasodilator tone, we have previously shown that NO bioactivity may be transported in blood, and have biological effects at a distance from the site of entry into the circulation. These endocrine effects of NO are mediated by intravascular NO-stores - candidates are protein and heme-bound NO species (RXNO) in plasma or erythrocytes and the oxidative NO-metabolite nitrite. Cumulating evidence suggests that nitrite may serve as a major intravascular storage pool for NO. Recent studies by our group show that regional, intra-arterial infusion of nitrite elicits downstream vasodilator response. The mechanism of nitrite reduction in vivo may involve a number of pathways. We have observed that nitrite is reduced to NO by its reaction with deoxyheme proteins. This chemistry suggests a role for hemoglobin and other heme proteins as an oxygen dependent nitrite reductase and further that nitrite ions might contribute to systemic hypoxic vasodilation. Other research groups have proposed pH-dependent mechanisms, the involvement of electron donors such as ascorbic acid, or xanthinoxidase as a reducing agent.

The present study will be conducted in two stages (Parts A and B) with the following objectives: Part A will determine 1) whether systemic (intravenous) infusion of nitrite modulates vascular tone in the systemic circulation, 2) whether oxypurinol (a potent inhibitor of xanthine oxidase activity) lowers or ascorbic acid potentiates nitrite-induced vasodilation, 3) elucidate the pharmacokinetic profile of nitrite application in humans and 4) determine phase I data for dosing nitrite in human disease. Part B will determine whether the systemic and pulmonary vascular responses to nitrite infusion are potentiated under hypoxic conditions and are mediated by NO gas per se as measured by NO content in exhaled breath.

ELIGIBILITY:
* ELIGIBILITY:

A total of 30 healthy volunteers will be enrolled in this study, 20 for Part A and 10 for Part B. All volunteer subjects will undergo screening with complete history, cardiovascular physical examination, blood collection for clinical chemistry routine analyses, plus testing for G-6-P-DH deficiency in erythrocytes and blood gas analysis via cooximetry, and a pregnancy test.

INCLUSION CRITERIA:

Subjects must be 21-40 years of age.

Subject must be in good health.

Subjects must provide informed, written consent for participation in this study.

Female subjects of childbearing age must have a negative pregnancy test.

EXCLUSION CRITERIA:

Subjects with a history or evidence of present or past hypertension (blood pressure greater than 140/90 mmHg), hypercholesterolemia (LDL cholesterol greater than 160 mg/dL), or diabetes mellitus (fasting blood glucose greater than 126 mg/dL)

Subjects who have a history of smoking within two years

Subjects who have a history of cardiovascular disease, peripheral vascular disease, coagulopathy, or any other disease predisposing to vasculitis or Raynaud's phenomenon.

Individuals with a future cardiovascular risk greater than 1 % in the next 10 years will be excluded from the study. Risk will be calculated using the Framingham risk calculator published on the web site: http://hin.nhlbi.nih.gov/atpiii/calculator.asp?usertype=prof.

Subjects with red blood cell G6PD deficiency (levels below the lower limits of normal).

Subjects with known cytochrome B5 deficiency will not participate in this study.

Subjects with a history of reaction to a medication or other substance characterized by dyspnea and cyanosis will not participate in this study.

Subjects with a baseline methemoglobin level greater than 1.9% will not receive nitrite infusions.

Lactating females will not participate since nitrite crosses into breast milk and could cause methemoglobinemia in the infant.

No volunteer subject will be allowed to take any medication (oral contraceptive agents are allowed), vitamin supplements that contain arginine, herbal preparations, nutriceuticals or other "alternative therapies" for at least one month prior to study and will not be allowed to take aspirin for one week prior to study

Subjects with a blood pressure of less than 90/60 mmHg or a MAP (mean arterial blood pressure) of less than 70 on the study day will be excluded from the protocol.

Due to exposure of high doses of ascorbic acid in this protocol calcium oxalate stone formers, patients on dialysis or with serious kidney disease, and patients with hemochromatosis and other iron overload diseases will be excluded.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2005-01-19; Study Completion 2011-04-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Boucher JL, Moali C, Tenu JP. Nitric oxide biosynthesis, nitric oxide synthase inhibitors and arginase competition for L-arginine utilization. Cell Mol Life Sci. 1999 Jul;55(8-9):1015-28. doi: 10.1007/s000180050352. PMID 10484661
- [Background] Furchgott RF, Zawadzki JV. The obligatory role of endothelial cells in the relaxation of arterial smooth muscle by acetylcholine. Nature. 1980 Nov 27;288(5789):373-6. doi: 10.1038/288373a0. PMID 6253831
- [Background] Ignarro LJ. Biosynthesis and metabolism of endothelium-derived nitric oxide. Annu Rev Pharmacol Toxicol. 1990;30:535-60. doi: 10.1146/annurev.pa.30.040190.002535. No abstract available. PMID 2188578